CLINICAL TRIAL: NCT05241925
Title: Effects of Continuous and Interval Physical Training Through the Intensity of the Incremental Shuttle Walk Test, on Functional Capacity and Quality of Life in Women With Malignant Breast Cancer During Chemotherapy Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, LUCIANA MARIA MALOSA SAMPAIO, PhD, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breast Cancer
Record Dates: First submitted 2022-01-26; First posted 2022-02-16 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer Female; Exercise Addiction
Keywords: Breast Cancer; Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined Training + Resistance Training (Experimental): Combined training (continuous aerobic + resistance) The protocol will consist of supervised exercise lasting 1h10min each session (5 min of warm-up, 30 min of aerobic exercise, 30 min of resistance exercise and 5 min of cool-down/relaxation).
  And Resistance Training
  - Resistance exercise will be performed at 70-80% of one repetition maximum (1-RM); 2 to 3 sets of 8 to 12 repetitions. The main muscle groups will be trained using training equipment with free weights and body mass of the participants. Exercises included leg extension, seated bicep curl, squat, seated triceps extension, sit-up, seated shoulder press, and standing pulldown
  Interventions: Other: Rehabilitation, exercise
- Hitt Training + Resistance Training (Experimental): Combined training (high-intensity interval (IAI) + resistance) - Supervised exercise lasting 30 min each session (5 min warm-up, 20 min IAI and 5 min cool-down/relaxation).
  And Resistance Training
  - Resistance exercise will be performed at 70-80% of one repetition maximum (1-RM); 2 to 3 sets of 8 to 12 repetitions. The main muscle groups will be trained using training equipment with free weights and body mass of the participants. Exercises included leg extension, seated bicep curl, squat, seated triceps extension, sit-up, seated shoulder press, and standing pulldown
  Interventions: Other: Rehabilitation, exercise

INTERVENTIONS:
Other: Rehabilitation, exercise — Combined training (continuous aerobic + resistance) The protocol will consist of supervised exercise lasting 1h10min each session (5 min of warm-up, 30 min of aerobic exercise, 30 min of resistance exercise and 5 min of cool-down/relaxation).
  Combined training (high-intensity interval (IAI) + resistance) - Supervised exercise lasting 30 min each session (5 min warm-up, 20 min IAI and 5 min cool-down/relaxation).
  And Resistance Training
  - Resistance exercise will be performed at 70-80% of one repetition maximum (1-RM); 2 to 3 sets of 8 to 12 repetitions. The main muscle groups will be trained using training equipment with free weights and body mass of the participants. Exercises included leg extension, seated bicep curl, squat, seated triceps extension, sit-up, seated shoulder press, and standing pulldown

SUMMARY:
Cancer on the world stage remains a major public health problem and the most common type among women.

Female breast cancer survivors often have multiple comorbidities such as diabetic, heart disease, sarcopenia, arthritis, hypertension, and others. In addition to fatigue, reduced functional capacity of the affected upper limb and decreased quality of life. The effects of antineoplastic treatment associated with chronic diseases predispose the emergence of cardiotoxicity, increasing the risk of developing cardiovascular diseases (CVD) and may lead to a decline in quality of life. This situation is due to the adverse effects that antineoplastic therapy exerts on the cardiovascular system.

According to the American Heart Association and American Cancer Society, physical exercise is one of the strategies adopted to prevent and reduce the effects of anticancer therapy, promoting effects on cardiovascular reserve5,6. Currently, although physical activity is essential for cancer survivors, the most effective exercise strategies (intensity, duration and type of exercise) to improve complications from breast cancer have not yet been defined.

The aim of the study is to investigate the effects of different types of physical training associated with functional capacity and quality of life in women undergoing antineoplastic treatment for breast cancer.

DETAILED DESCRIPTION:
Cancer is a universal term used for a large group of diseases, characterized by the disordered growth of cells beyond their usual limits, which can affect adjacent parts of the body and/or spread to other organs and tissues. Breast cancer worldwide is a major public health problem, being among all types of neoplasm the most common among women, regardless of age and ethnicity.

Treatment for breast cancer may include surgery, radiation therapy, and systemic therapies such as chemotherapy, hormone therapy, or biological therapy. A number of factors are considered to determine the treatment and sequence of therapies. With advances in early detection and treatment of cancer, the survival rate has increased in more developed countries, reaching 85% in the first five years after diagnosis.

The survival of patients with breast cancer has increased, generating greater concern for the individual's overall well-being. Chemotherapy treatments can cause short or long-term cardiorespiratory limitations, reduced functional capacity and worse quality of life, making daily activities difficult for these patients.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of confirmed breast cancer. Duration of adjuvant chemotherapy treatment. Undergoing surgery for breast cancer treatment.

Exclusion Criteria:

* neoplasm prior to breast cancer
* heart disease;
* musculoskeletal disorder;
* respiratory disease;
* uncontrolled arterial hypertension - factors that limit the performance of any of the assessments and/or training in the study.
* Not having undergone chemotherapy or radiotherapy prior to the diagnosis of breast cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Distance Incremental Shuttle Walk Test (SWTI) | Distance Incremental Shuttle Walk Test (SWTI)
  Distance walking meters
Maximum endurance test (1RM) | Maximum endurance test (1RM)
  Kg

SECONDARY OUTCOMES:
Time Grocery Shelving Task Test | Time Grocery Shelving Task Test
  Seconds
European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30) | European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30)
  Score
Functional Assessment of Breast Cancer Therapy Questionnaire (FACT-B) | Functional Assessment of Breast Cancer Therapy Questionnaire (FACT-B)
  Score
Brief Fatigue Inventory Questionnaire (BFI) | Brief Fatigue Inventory Questionnaire (BFI)
  Score

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Sampaio, PhD, Principal Investigator — University of Nove de Julho

IPD SHARING:
Plan to Share IPD: No